CLINICAL TRIAL: NCT04474132
Title: Feasibility Study for Finger Prick Testing of Presence of Current and or Previous T. Gondii Infection
Brief Title: Point of Care Testing for Presence of Current and or Previous T. Gondii Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB20-0442
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Toxoplasma Infections
Keywords: toxoplasma; test; feasibility

STUDY DESIGN:
Intervention Model Description: subjects are recruited continuously and being tested with the study device as well as with the standard cleared test for the presence of Toxoplasma gondii antibody.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- single group (Other): binary: positive or negative result
  Interventions: Device: toxoplasma ICT IgG-IgM BK

INTERVENTIONS:
Device: toxoplasma ICT IgG-IgM BK — a point-of-care device, using blood from finger stick to measure the presence or absence of anti Toxoplasma gondii antibody

SUMMARY:
This is part of a feasibility study to compare the predicate standard FDA cleared test for serum to a point of care test Toxoplasma ICT IgG-IgM BK produced by LD Bio Diagnostic. The specificity and sensitivity in testing serum and whole blood will be compared. This study includes 70 persons either pregnant or non pregnant.

This is being done in accordance with FDA requirements for clearance of a testing device . The investigators will use a standard FDA cleared test in all studies. The FDA has suggested that the investigators submit a pre subQ for a 510K and dual CLIA waiver.

This allows the investigators also to determine feasibility of use of the predicate test in conjunction with the experimental test with volunteers, including men, women, and pregnant women.

DETAILED DESCRIPTION:
This study will determine the feasibility of using the point of care Toxoplasma ICT IgG-IgM BK test produced by LD Bio Diagnostic to detect Toxoplasma gondii in clinical settings. The result of testing from Toxoplasma ICT IgG-IgM BK test will be compared with the standard predicate test. These results will be provided to FDA for consideration for clearance of this test.

ELIGIBILITY:
Inclusion Criteria:

* any adult who is willing to participate in the study

Exclusion Criteria:

* pregnant women who are in their 17-27 weeks of gestation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
congruence of Toxoplasma ICT IgG-IgM test and standard predicate test | two weeks for initial result and a year for whole study
  Toxoplasma ICT IgG-IgM test is feasible and the test result of the study device is same with the result of standard cleared test

CONTACTS AND LOCATIONS:
Overall Officials: Rima McLeod, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lykins J, Li X, Levigne P, Zhou Y, El Bissati K, Clouser F, Wallon M, Morel F, Leahy K, El Mansouri B, Siddiqui M, Leong N, Michalowski M, Irwin E, Goodall P, Ismail M, Christmas M, Adlaoui EB, Rhajaoui M, Barkat A, Cong H, Begeman IJ, Lai BS, Contopoulos-Ioannidis DG, Montoya JG, Maldonado Y, Ramirez R, Press C, Peyron F, McLeod R. Rapid, inexpensive, fingerstick, whole-blood, sensitive, specific, point-of-care test for anti-Toxoplasma antibodies. PLoS Negl Trop Dis. 2018 Aug 16;12(8):e0006536. doi: 10.1371/journal.pntd.0006536. eCollection 2018 Aug. No abstract available. PMID 30114251
- [Result] Begeman IJ, Lykins J, Zhou Y, Lai BS, Levigne P, El Bissati K, Boyer K, Withers S, Clouser F, Noble AG, Rabiah P, Swisher CN, Heydemann PT, Contopoulos-Ioannidis DG, Montoya JG, Maldonado Y, Ramirez R, Press C, Stillwaggon E, Peyron F, McLeod R. Point-of-care testing for Toxoplasma gondii IgG/IgM using Toxoplasma ICT IgG-IgM test with sera from the United States and implications for developing countries. PLoS Negl Trop Dis. 2017 Jun 26;11(6):e0005670. doi: 10.1371/journal.pntd.0005670. eCollection 2017 Jun. PMID 28650970
- [Result] Gomez CA, Budvytyte LN, Press C, Zhou L, McLeod R, Maldonado Y, Montoya JG, Contopoulos-Ioannidis DG. Evaluation of Three Point-of-Care Tests for Detection of Toxoplasma Immunoglobulin IgG and IgM in the United States: Proof of Concept and Challenges. Open Forum Infect Dis. 2018 Oct 29;5(10):ofy215. doi: 10.1093/ofid/ofy215. eCollection 2018 Oct. PMID 30393749
- [Derived] Zhou Y, Leahy K, Grose A, Lykins J, Siddiqui M, Leong N, Goodall P, Withers S, Ashi K, Schrantz S, Tesic V, Abeleda AP, Beavis K, Clouser F, Ismail M, Christmas M, Piarroux R, Limonne D, Chapey E, Abraham S, Baird I, Thibodeau J, Boyer KM, Torres E, Conrey S, Wang K, Staat MA, Back N, L'Ollivier C, Mahinc C, Flori P, Gomez-Marin J, Peyron F, Houze S, Wallon M, McLeod R. Novel paradigm enables accurate monthly gestational screening to prevent congenital toxoplasmosis and more. PLoS Negl Trop Dis. 2024 May 28;18(5):e0011335. doi: 10.1371/journal.pntd.0011335. eCollection 2024 May. PMID 38805559